CLINICAL TRIAL: NCT01951118
Title: Olfactory Deficits and Donepezil Treatment in Cognitively Impaired Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Davangere P. Devanand, Professor of Clinical Psychiatry and Neurology, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6655; 1R01AG041795 (NIH)
Record Dates: First submitted 2013-09-18; First posted 2013-09-26 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Delirium, Dementia, Amnestic, Cognitive Disorders
Keywords: Smell; Olfaction Disorders; Atropine; Donepezil; Cholinesterase Inhibitors; Cognition Disorders
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Neurocognitive Disorders; Anosmia; Olfaction Disorders; Cognition Disorders | interventions — Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Donepezil Treatment & Atropine Challenge (Experimental): Atropine nasal spray is administered at baseline for the atropine challenge which involves administration of the 40-item UPSIT immediately before and 45 minutes after atropine administration. Immediately after the atropine challenge, donepezil treatment is started and continues for 52 weeks.
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Donepezil — Donepezil 5mg will be given for 4 weeks and if tolerated, the dose will be increased to 10 mg per day. The dose range of 5 to 10 mg of donepezil per day will be continued for the study duration, and this is the recommended dose for donepezil in the treatment of mild to moderate Alzheimer's disease. For patients who do not tolerate donepezil or have a history of intolerance to donepezil or cannot take donepezil for other reasons, treatment with other cholinesterase inhibitors (galantamine or rivastigmine) is permitted at any stage of the protocol. Data will be analyzed in two ways: for donepezil alone, and for any cholinesterase inhibitor (donepezil or rivastigmine or galantamine) as the intervention.
  Other Names: Aricept

SUMMARY:
Olfactory identification deficits occur in patients with Alzheimer's disease (AD), are associated with disease severity, predict conversion from mild cognitive impairment (MCI) to AD and are associated with healthy elderly subjects developing MCI. Odor (olfactory) identification deficits may reflect degeneration of cholinergic inputs to the olfactory bulb and other olfactory brain regions. Acetylcholinesterase inhibitors (ACheI) like donepezil show modest effects in improving cognition but can be associated with adverse effects and increased burden and costs because of the need for prolonged, often lifelong, treatment. Converging findings on odor identification test performance (UPSIT, scratch and sniff 40-item test) from four pilot studies, including two of our own, suggest that acute change in the UPSIT in response to an anticholinergic challenge (atropine nasal spray), incremental change over 8 weeks, and even the baseline UPSIT score by itself, may predict cognitive improvement with ACheI treatment in MCI and AD. If change in odor identification deficits can help to identify which patients should receive ACheI treatment, this simple inexpensive approach will advance the goal of improving personalized treatment, improve selection and monitoring of patients for ACheI treatment, reduce needless ACheI exposure with risk of side effects, and decrease health care costs.

DETAILED DESCRIPTION:
In this clinical trial, the investigators will evaluate, treat and follow two broad samples of adult patients at New York State Psychiatric Institute/Columbia University Medical Center. Study 1 will include 70 patients with amnestic Mild Cognitive Impairment (MCI). Study 2 will include 100 patients with probable Alzheimer's Disease (AD). Recruitment will be from clinics and/or advertisements. In the protocol, all 170 patients will receive baseline memory and olfactory assessments and are treated with donepezil. Patients will be followed for a total of 1 year. During this time, patients will be monitored closely by the study physician and will receive memory and olfactory assessments at weeks 0, 8, 26, and 52. In addition, an olfactory challenge test will be done at baseline.

This project will be of value in the selection of patients with MCI and AD for treatment based on the evaluation of olfaction tests to predict response to donepezil. Since mild cognitive impairment is widespread and Alzheimer's disease represents a major public health problem, this study has considerable public purpose and significance.

ELIGIBILITY:
Study 1

Inclusion Criteria:

* Of either sex, age 55-95 years old
* Patients who meet criteria for amnestic mild cognitive impairment by meeting all of the following:

  (i) subjective memory complaints (ii) Wechsler Memory Scale-III Logical Memory combined Story A + B immediate recall score or combined Story A + B delayed recall score or Free and Cued Selective Reminding Test immediate recall or delayed recall score greater than 1.5 Standard Deviation (SD) below norms or Selective Reminding Test immediate recall or delayed recall score greater than 1.5 SD below norms iii) no functional impairment consistent with dementia
* Folstein Mini Mental State (MMSE) score ≥ 23 out of 30
* Clinical Dementia Rating (CDR) of 0.5 (questionable dementia)
* Availability of informant
* Retains capacity to consent

Exclusion Criteria:

* Medical contraindication to donepezil treatment or prior history of intolerability to donepezil treatment.
* Medications with anticholinergic effects that have been shown to adversely impact cognition will not be permitted. Benzodiazepines in lorazepam equivalents less than or equal to 2 mg daily and narcotics will also not be permitted.
* Meets criteria for dementia by Diagnostic and Statistical Manual IV (DSM-IV) or probable Alzheimer's disease by National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA)
* Meets Diagnostic and Statistical Manual IV Text Revision (DSM IV TR) criteria for: (i)schizophrenia, schizoaffective disorder, other psychosis, or bipolar I disorder (ii)alcohol or substance dependence or abuse (current or within past 6 months)
* Current untreated major depression or suicidality
* Parkinson's disease, Lewy body disease, multiple sclerosis, central nervous system infection, Huntington's disease, amyotrophic lateral sclerosis, other major neurological disorder.
* Mental Retardation
* Cystic Fibrosis
* Clinical stroke with residual neurological deficits. MRI findings of cerebrovascular disease (small infarcts, lacunes, periventricular disease) in the absence of clinical stroke with residual neurological deficits will not lead to exclusion.
* Patients receiving cholinesterase inhibitors (donepezil, rivastigmine, galantamine) or memantine will be excluded. Patients already receiving one of these medications at screening who undergo a 2-week washout before starting all study procedures will not be excluded.
* Acute, severe, unstable medical illness. For cancer, patients with active illness or metastases will be excluded, but past history of successfully treated cancer will not lead to exclusion.
* Exclusion criterion for olfaction: history of anosmia due to any cause (e.g. traumatic or congenital) verified by UPSIT score of <11 out of 40; head trauma with loss of consciousness; nasal sinus disease, current upper respiratory infection; severe allergies to odors; current smoker > 1 pack daily.
* Exclusion criteria for atropine nasal spray: presence of nasal deformity or disease that makes it difficult to administer the nasal spray reliably. A patient who cannot complete the atropine nasal spray procedure can still participate in the rest of the study.

Study 2

Inclusion Criteria:

* Of either sex, age 55-95 years old
* Diagnosis of probable Alzheimer's disease (NINCDS-ADRDA criteria) and the diagnosis of "Probable AD dementia: core clinical diagnosis with amnestic or nonamnestic initial presentation".
* Folstein Mini Mental State (MMSE) score 18-27 out of 30
* Availability of informant
* Retains capacity to consent

Exclusion Criteria:

* Medical contraindication to donepezil treatment or prior history of intolerability to donepezil treatment.
* Medications with anticholinergic effects that have been shown to adversely impact cognition will not be permitted. Benzodiazepines in lorazepam equivalents less than or equal to 2 mg daily and narcotics will also not be permitted.
* Meets DSM IV TR criteria for:(i)schizophrenia, schizoaffective disorder, other psychosis, or bipolar I disorder (ii)alcohol or substance dependence or abuse (current or within past 6 months)
* Current untreated major depression or suicidality
* Parkinson's disease, Lewy body disease, multiple sclerosis, central nervous system infection, Huntington's disease, amyotrophic lateral sclerosis, other major neurological disorder.
* Mental Retardation
* Cystic Fibrosis
* Clinical stroke with residual neurological deficits. MRI findings of cerebrovascular disease (small infarcts, lacunes, periventricular disease) in the absence of clinical stroke with residual neurological deficits will not lead to exclusion.
* Patients receiving cholinesterase inhibitors (donepezil, rivastigmine, galantamine) or memantine will be excluded. Patients already receiving one of these medications at screening who undergo a 2-week washout before starting all study procedures will not be excluded.
* Acute, severe, unstable medical illness. For cancer, patients with active illness or metastases will be excluded, but past history of successfully treated cancer will not lead to exclusion.
* Exclusion criterion for olfaction: history of anosmia due to any cause (e.g. traumatic or congenital) verified by UPSIT score of <11 out of 40; head trauma with loss of consciousness; nasal sinus disease, current upper respiratory infection; severe allergies to odors; current smoker > 1 pack daily.
* Exclusion criteria for atropine nasal spray: presence of nasal deformity or disease that makes it difficult to administer the nasal spray reliably. A patient who cannot complete the atropine nasal spray procedure can still participate in the rest of the study.

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davangere Devanand, M.D., Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- [Derived] Devanand DP, Liu X, Chunga RE, Cohen H, Andrews H, Schofield PW, Stern Y, Huey ED, Choi J, Pelton GH. Odor Identification Impairment and Change with Cholinesterase Inhibitor Treatment in Mild Cognitive Impairment. J Alzheimers Dis. 2020;75(3):845-854. doi: 10.3233/JAD-200021. PMID 32333591

RESULTS

PARTICIPANT FLOW:
Groups:
- Donepezil Treatment & Atropine Challenge: Atropine nasal spray is administered at baseline for the atropine challenge which involves administration of the 40-item UPSIT immediately before and 45 minutes after atropine administration. Immediately after the atropine challenge, donepezil treatment is started and continues for 52 weeks.
  Donepezil: Donepezil 5mg will be given for 4 weeks and if tolerated, the dose will be increased to 10 mg per day. The dose range of 5 to 10 mg of donepezil per day will be continued for the study duration, and this is the recommended dose for donepezil in the treatment of mild to moderate Alzheimer's disease. For patients who do not tolerate donepezil or have a history of intolerance to donepezil or cannot take donepezil for other reasons, treatment with other cholinesterase inhibitors (galantamine or rivastigmine) is permitted at any stage of the protocol. Data will be analyzed in two ways: for donepezil alone, and for any cholinesterase inhibitor (donepezil or rivastigmine or galantamine).
Period: Overall Study
Arm/Group | Donepezil Treatment & Atropine Challenge
Started | 121
Completed | 94
Not Completed | 27

BASELINE CHARACTERISTICS:
Arm/Group | Donepezil Treatment & Atropine Challenge
Number analyzed (Participants) | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 81
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21
  Not Hispanic or Latino | 100
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 27
  White | 88
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 121

OUTCOME MEASURES:

1. Primary Outcome: Change Over Time in Selective Reminding Test (SRT) Scores
Description: The Selective Reminding Test (SRT) is a 12-item test of verbal learning and memory. To administer, the researcher will read aloud a list of 12 words. The participant repeats each word aloud to ensure that the word was heard correctly. Immediately following the reading of all 12 words, the participant is asked to recall as many words as possible within the one minute time limit. The participant is then reminded of the words they did not say and asked to recall the list again. This process is repeated for 6 trials. The total immediate recall is the total number of words recalled by the participant from all 6 trials. This is the number that is reported. Lower scores indicate fewer words recalled and a poorer performance.
Time Frame: Week 0, Week 8, Week 26, Week 52
Population: The number analyzed in one or more rows differs from overall number analyzed due to participant drop-out.
Measure: Mean (Standard Deviation); unit: Words
Groups:
- MCI Sample: 100 patients with MCI were analyzed for this sample.
- AD Sample: 21 patients with AD were analyzed for this sample.
Arm/Group | MCI Sample | AD Sample
Number analyzed (Participants) | 100 | 21
Words
  Week 0 | 36.14 (10.67) | 21.19 (8.23)
  Week 8: number analyzed (Participants) | 90 | 20
  Week 8 | 39.99 (10.30) | 24.10 (9.82)
  Week 26: number analyzed (Participants) | 83 | 20
  Week 26 | 39.75 (10.69) | 23.00 (8.07)
  Week 52: number analyzed (Participants) | 77 | 16
  Week 52 | 39.62 (11.44) | 24.38 (9.69)

2. Secondary Outcome: Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog)
Description: The modified Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog) is a cognitive battery that assesses learning, memory, language production, language comprehension, constructional praxis, ideational praxis, and orientation. The ADAS-Cog is not a timed test and the participant's score does not depend on how rapidly the test is completed. The ADAS-Cog total score is based on the total number of errors made in the test by the participant. Therefore, a lower total score indicates a higher cognitive performance. The total score ranges from 0 to 95 and is determined by summing the errors from 12 subscales. The total score, indicating number of errors made, is the number that is reported at each timeframe.
Time Frame: Week 0, Week 8, Week 26, Week 52
Population: The number analyzed in one or more rows differs from overall number analyzed due to participant drop-out.
Measure: Mean (Standard Deviation); unit: Errors
Groups:
- MCI Sample: 100 MCI participants were analyzed for this sample.
- AD Sample: 21 AD participants were analyzed for this sample.
Arm/Group | MCI Sample | AD Sample
Number analyzed (Participants) | 100 | 21
Errors
  Week 0: number analyzed (Participants) | 99 | 21
  Week 0 | 11.41 (4.67) | 21.67 (6.12)
  Week 8: number analyzed (Participants) | 89 | 20
  Week 8 | 10.13 (4.22) | 19.30 (5.80)
  Week 26: number analyzed (Participants) | 83 | 20
  Week 26 | 9.63 (4.44) | 19.63 (7.15)
  Week 52: number analyzed (Participants) | 77 | 15
  Week 52 | 10.40 (4.72) | 22.69 (8.99)

3. Secondary Outcome: Clinician's Interview Based Impression (CIBIC-plus)
Description: The CIBIC-plus is a well-validated, reliable and widely used measure (range 1-7) of global improvement used in AD and MCI trials. This is a measure of change based on clinician impression. Higher values represent a worse outcome.
Time Frame: Week 8, Week 26, Week 52
Population: The number analyzed in one or more rows differs from overall number analyzed due to participant drop-out.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI Sample | AD Sample
Number analyzed (Participants) | 100 | 21
units on a scale
  Week 8: number analyzed (Participants) | 89 | 20
  Week 8 | 3.34 (0.74) | 3.55 (0.69)
  Week 26: number analyzed (Participants) | 82 | 20
  Week 26 | 3.15 (0.86) | 3.75 (0.64)
  Week 52: number analyzed (Participants) | 76 | 16
  Week 52 | 3.11 (1.17) | 4.38 (0.96)

4. Secondary Outcome: Pfeffer Functional Activities Questionnaire (FAQ)
Description: FAQ is a widely used 10-item instrument that takes 3 minutes to administer and focuses on instrumental, social and cognitive functioning. The assessment is completed by a study informant - typically a caregiver able to report best on the patient's current ability. The instrument assesses the patient's current ability, at the point of testing and through the past month, in these various domains. The total score is described as the cumulative scores of each item, ranging from "0 - No help needed" to "3 - No, unable to do." More impairment is indicated by higher scores. The reported total score range is from 0 (no impairment score) to 30 (maximum impairment score).
Time Frame: Week 0, Week 8, Week 26, Week 52
Population: The number analyzed in one or more rows differs from overall number analyzed due to participant drop-out.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI Sample | AD Sample
Number analyzed (Participants) | 100 | 21
units on a scale
  Week 0: number analyzed (Participants) | 94 | 16
  Week 0 | 4.80 (4.84) | 11.25 (6.19)
  Week 8: number analyzed (Participants) | 83 | 18
  Week 8 | 4.68 (4.56) | 11.78 (4.72)
  Week 26: number analyzed (Participants) | 77 | 20
  Week 26 | 4.84 (4.96) | 13.75 (5.46)
  Week 52: number analyzed (Participants) | 74 | 13
  Week 52 | 4.25 (4.76) | 14.62 (4.15)

5. Secondary Outcome: Measurement of Everyday Cognition (Ecog)
Description: This instrument has 40 items, takes 20 minutes to administer, and focuses on functional correlates of cognitive deficits. This assessment asks the study informant to rate the participant's ability to perform certain tasks with the domains of Memory, Language, Visual-spatial and Perceptual Abilities, Executive Functioning: Planning, Executive Functioning: Organization, and Executive Functioning: Divided Attention. The informant is asked to compare functioning from 10 years prior to the time of testing. The Everyday Cognition measure uses the sum score of all of the subscales, and the items are reverse coded (i.e., 1= "Better or no change", 2="Questionable/occasionally worse", 3="Consistently a little worse", 4="Consistently much worse"), meaning that lower scores are better. Reported total scores range from 39 (Better or no change) to 156 (Consistently much worse).
Time Frame: Week 0, Week 8, Week 26, Week 52
Population: The number analyzed in one or more rows differs from overall number analyzed due to participant drop-out.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- MCI Sample: 100 MCI participants were included in this sample.
- AD Sample: 21 AD participants were included in this sample.
Arm/Group | MCI Sample | AD Sample
Number analyzed (Participants) | 100 | 21
units on a scale
  Week 0: number analyzed (Participants) | 92 | 20
  Week 0 | 67.93 (20.58) | 90.80 (28.11)
  Week 8: number analyzed (Participants) | 83 | 20
  Week 8 | 67.88 (23.35) | 89.20 (31.14)
  Week 26: number analyzed (Participants) | 77 | 20
  Week 26 | 67.92 (23.20) | 97.65 (29.02)
  Week 52: number analyzed (Participants) | 74 | 17
  Week 52 | 66.84 (22.66) | 103.59 (29.27)

6. Other Pre Specified Outcome: Mini-Mental State Examination - MMSE
Description: The Mini Mental State Examination (MMSE) is a widely used 30-item test of cognitive function that includes tests of orientation, attention, memory, language, and visual-spatial skills. Values range from 0-30; a higher value represents a better outcome.
Time Frame: Week 0, Week 26, Week 52
Population: The number analyzed in one or more rows differs from overall number analyzed due to participant drop-out.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI Sample | AD Sample
Number analyzed (Participants) | 100 | 21
units on a scale
  Week 0 | 26.72 (2.17) | 23.048 (2.40)
  Week 26: number analyzed (Participants) | 83 | 20
  Week 26 | 26.90 (2.20) | 21.20 (3.52)
  Week 52: number analyzed (Participants) | 77 | 17
  Week 52 | 26.44 (2.47) | 20.35 (3.71)

7. Other Pre Specified Outcome: Trail Making Test (Parts A and B)
Description: Parts A and B are composed of 25 circles. Patients are asked to scan the entire page and identify the next number or letter in a sequence.
Time Frame: Week 0, Week 52
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Wechsler Adult Intelligence Scale (WAIS) -III Digit Symbol Subtest
Description: The Wechsler Adult Intelligence Scale (WAIS) -III Digit Symbol Subtest is a paper-and-pencil cognitive test presented on a single sheet of paper that requires a subject to match symbols to numbers according to a key located on the top of the page. Values range from 0-93; a higher value represents a better outcome.
Time Frame: Week 0, Week 52
Population: The number analyzed in one or more rows differs from overall number analyzed due to participant drop-out.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI Sample | AD Sample
Number analyzed (Participants) | 100 | 21
units on a scale
  Week 0: number analyzed (Participants) | 99 | 19
  Week 0 | 36.83 (13.72) | 25.47 (9.27)
  Week 52: number analyzed (Participants) | 76 | 16
  Week 52 | 37.24 (12.17) | 21.06 (11.66)

9. Other Pre Specified Outcome: Controlled Word Association (CFL)
Time Frame: Week 0, Week 52
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Boston Naming Test (BNT)
Time Frame: Week 0, Week 52
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Wechsler Memory Scale (WMS)-R Digit Span
Time Frame: Week 0, Week 52.
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Treatment Emergent Symptom Scale (TESS)
Description: The Treatment Emergent Symptom Scale (TESS) is widely used to evaluate somatic side effects. For each item, a rating is made on a 3-point scale, with an additional rating on the likelihood that the medication caused the side effect. Values range from 0-78; a higher value indicates a worse outcome.
Time Frame: Week 0, Week 8, Week 26, Week 52
Population: The number analyzed in one or more rows differs from overall number analyzed due to participant drop-out.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI Sample | AD Sample
Number analyzed (Participants) | 100 | 21
units on a scale
  Week 0: number analyzed (Participants) | 98 | 18
  Week 0 | 2.57 (2.62) | 1.89 (2.05)
  Week 8: number analyzed (Participants) | 88 | 17
  Week 8 | 1.61 (1.90) | 1.53 (1.37)
  Week 26: number analyzed (Participants) | 77 | 20
  Week 26 | 1.42 (1.86) | 1.20 (1.47)
  Week 52: number analyzed (Participants) | 74 | 16
  Week 52 | 1.28 (2.11) | 1.69 (2.33)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected beginning at study start through study conclusion, an average of 5 years.
Arm/Group | Donepezil Treatment & Atropine Challenge
All-Cause Mortality (participants affected / at risk) | 3/121
Serious Adverse Events (participants affected / at risk) | 8/121
Other Adverse Events (participants affected / at risk) | 0/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Donepezil Treatment & Atropine Challenge (N=121)
Low platelet level (Blood and lymphatic system disorders) | 1
Broken Femur (Musculoskeletal and connective tissue disorders) | 1
Agitation (Psychiatric disorders) | 1
Dizziness (General disorders) | 1
Wrist Fracture (Musculoskeletal and connective tissue disorders) | 1
Death (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-08-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT01951118/Prot_000.pdf
  • Statistical Analysis Plan (2012-03-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT01951118/SAP_001.pdf